CLINICAL TRIAL: NCT06925477
Title: Direct Selective Laser Trabeculoplasty (DSLT) and Selective Laser Trabeculoplasty (SLT) in Reducing Intraocular Pressure in Open-Angle Glaucoma
Brief Title: Direct vs. Conventional SLT in Open-Angle Glaucoma: A RCT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00142923
Record Dates: First submitted 2025-04-06; First posted 2025-04-13 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: GLAUCOMA 1, OPEN ANGLE, D (Disorder)
Keywords: Open Angle Glaucoma; SLT; Trabeculoplasty; DSLT
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm 1- DSLT (Direct Selective Laser Trabeculoplasty) (Other): DSLT is a well-established non-contact laser application that does not require a gonioscopy lens, reducing the risk of corneal damage and inflammation.
  Interventions: Device: DSLT treatment for Open-Angle Glaucoma
- Arm 2- Selective Laser Trabeculoplasty (SLT) (Other): SLT is a widely used and effective laser therapy to lower intraocular pressure that requires operator expertise and carries risks of mild inflammation, corneal damage and discomfort. This is a standard laser system that requires the use of a gonioscopy lens placed on the cornea to administer.
  Interventions: Device: SLT treatment for Open-Angle Glaucoma

INTERVENTIONS:
Device: DSLT treatment for Open-Angle Glaucoma — This intervention aims to determine the efficacy and safety of Direct Selective Laser Trabeculoplasty (DSLT) in reducing intraocular pressure in patients with open-angle glaucoma.
  Arms: Arm 1- DSLT (Direct Selective Laser Trabeculoplasty)
Device: SLT treatment for Open-Angle Glaucoma — To determine the efficacy and safety of using Selective Laser Trabeculoplasty for treatment of open-angle glaucoma.
  Arms: Arm 2- Selective Laser Trabeculoplasty (SLT)

SUMMARY:
This study compares two laser treatments for open-angle glaucoma: Selective Laser Trabeculoplasty (SLT) and Direct Selective Laser Trabeculoplasty (DSLT). SLT is a widely used procedure that requires a manual technique with a goniolens, while DSLT is a new, automated, non-contact method using the Eagle system. The study will evaluate whether DSLT is as effective as SLT in reducing intraocular pressure (IOP). Participants will be randomly assigned to receive either treatment and will be monitored over 12 months to assess changes in IOP, medication use, and safety outcomes. The goal is to determine if the simpler DSLT procedure can provide similar results to SLT, potentially improving patient comfort and access to glaucoma care.

DETAILED DESCRIPTION:
Glaucoma management is fundamentally aimed at reducing intraocular pressure (IOP) to prevent optic nerve damage and preserve vision. Selective Laser Trabeculoplasty (SLT) has been a cornerstone in the treatment of open-angle glaucoma due to its efficacy and safety profile. However, SLT's manual delivery method using a goniolens can introduce variability, patient discomfort, and operator dependency.

Direct Selective Laser Trabeculoplasty (DSLT) represents an innovative advancement, offering a non-contact, automated laser treatment via the Eagle system. This technology is designed to simplify the procedure, enhance patient comfort, and minimize operator-induced variability. Early evidence suggests that DSLT may provide similar or improved IOP reduction compared to SLT, with a potentially better safety profile.

This study seeks to rigorously evaluate whether DSLT is non-inferior to SLT in reducing IOP, thus providing critical data on the efficacy and safety of this novel approach. Demonstrating non-inferiority would support broader adoption of DSLT, potentially improving patient outcomes and expanding access to effective glaucoma treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Diagnosed with OAG (including exfoliative/pigmentary glaucoma) or OHT.
* Gonioscopically visible scleral spur for 360 degrees.
* Ability to provide informed consent.
* In good health, without prior laser trabeculoplasty, with decision to treat made by an ophthalmologist on the basis of risk profile, patient preference, or both.
* Each eye with one of the following qualifying diagnoses (diagnoses may differ between eyes):

  * High-risk ocular hypertension (OHT): IOP > 21 mmHg without glaucomatous optic neuropathy (excavation, diffuse or focal thinning or notching of the neuroretinal rim, visible nerve fiber layer defects, or asymmetry of the vertical cup-to-disc ratio of >0.2 between eyes) [enrollment of trial participants with High-risk OHT will be capped at 25% of total enrollment]
  * Mild primary open-angle glaucoma: glaucomatous optic neuropathy, visual field mean deviation >-6.0 dB with no points in the central 5° <15 dB
  * Moderate primary open-angle glaucoma: glaucomatous optic neuropathy, visual field mean deviation -6.0 dB to >-12 dB and no more than 1 central 5° point <15 dB

Exclusion Criteria:

* Advanced POAG in either eye
* Glaucoma other than OAG (including pigmentary and pseudoexfoliation glaucoma) in either eye
* Mean IOP > 35 mmHg at either the screening or baseline visit in either eye
* Narrow or closed angle (Shaffer Grade 0, 1, or 2) in either eye
* Contraindications to SLT, brimonidine, apraclonidine, or any other study intervention
* Any corneal pathology that would preclude accurate assessment of IOP by Goldmann tonometry in either eye
* Any intraocular surgical procedure within the past 6 months in either eye
* Inability to attend all scheduled study visits
* Pregnancy or plan to become pregnant in the next 1 year
* Any prior laser trabeculoplasty, including ALT, MLT and SLT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 6 months
  Measuring the difference in the average IOP measurement reduction from the patient's baseline at 6 months between the DSLT and the SLT groups.

SECONDARY OUTCOMES:
Secondary Outcome | 12 months
  The patients percentage of IOP reduction at 2 months, 6 months, and 12 months. Measuring the amount of patient's that have achieved >/= 20% IOP reduction at 6 months. Documentation of any change in the use of ocular hypotensive medications at 12 months. Documentation of the rate of repeat laser treatments or additional IOP lowering procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Jella An, MD, MBA, Principal Investigator — Medical University of South Carolina
Locations (1):
- MUSC Health West Ophthalmology Clinic, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Konstantakopoulou E, Gazzard G, Garway-Heath D, Adeleke M, Ambler G, Vickerstaff V, Bunce C, Nathwani N, Barton K; LiGHT Trial Study Group. Selective Laser Trabeculoplasty After Medical Treatment for Glaucoma or Ocular Hypertension. JAMA Ophthalmol. 2025 Apr 1;143(4):295-302. doi: 10.1001/jamaophthalmol.2024.6492. PMID 39976961
- [Result] Goldenfeld M, Belkin M, Dobkin-Bekman M, Sacks Z, Blum Meirovitch S, Geffen N, Leshno A, Skaat A. Automated Direct Selective Laser Trabeculoplasty: First Prospective Clinical Trial. Transl Vis Sci Technol. 2021 Mar 1;10(3):5. doi: 10.1167/tvst.10.3.5. PMID 34003939
- [Result] Melik Parsadaniantz S, Reaux-le Goazigo A, Sapienza A, Habas C, Baudouin C. Glaucoma: A Degenerative Optic Neuropathy Related to Neuroinflammation? Cells. 2020 Feb 25;9(3):535. doi: 10.3390/cells9030535. PMID 32106630